CLINICAL TRIAL: NCT06745102
Title: Effect of Iso-alpha Acids and Xanthohumol on the Human Immune System in Overweight People With the Onset of Metabolic Diseases
Brief Title: Hop Compounds on the Immune System in Overweight People
Acronym: ÜG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ina Bergheim, Principal Investigator, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UVienna24
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Response
MeSH Terms: interventions — xanthohumol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Xanthohumol (Experimental): Participants receive a study drink supplemented with Xanthohumol (0 mg = Placebo or 0.75 mg soluble Xanthohumol)
  Interventions: Dietary Supplement: Xanthohumol
- Iso-alpha Acids (Experimental): Participants receive a study drink supplemented with Iso-alpha Acids (0 mg = Placebo or 45 mg Iso-alpha Acids)
  Interventions: Dietary Supplement: Iso-alpha Acids
- Xanthohumol + Iso-alpha Acids (Experimental): Participants receive a study drink supplemented with Xanthohumol + Iso-alpha Acids (0 mg = Placebo or 0.75 mg + 45 mg soluble Xanthohumol + Iso-alpha Acids)
  Interventions: Dietary Supplement: Xanthohumol + Iso-alpha Acids

INTERVENTIONS:
Dietary Supplement: Xanthohumol — Participants receive a study drink supplemented with Xanthohumol (0 mg = Placebo or 0.75 mg soluble Xanthohumol)
  Arms: Xanthohumol
Dietary Supplement: Iso-alpha Acids — Participants receive a study drink supplemented with Iso-alpha Acids (0 mg = Placebo or 45 mg Iso-alpha Acids)
  Arms: Iso-alpha Acids
Dietary Supplement: Xanthohumol + Iso-alpha Acids — Participants receive a study drink supplemented with Xanthohumol and Iso-alpha Acids (0 mg = Placebo or 0.75 mg + 45 mg soluble Xanthohumol + Iso-alpha Acids)
  Arms: Xanthohumol + Iso-alpha Acids

SUMMARY:
The aim of the present study is to determine the effect of Iso-alpha Acids and Xanthohumol from hops on the immune response in overweight participants.

DETAILED DESCRIPTION:
The aim of the present study is to investigate whether the oral intake of Xanthohumol and Iso-alpha Acids has different protective effects on the immune response of isolated blood cells from overweight people with people with incipient metabolic diseases, what the time course of the effect is and whether the levels of the substances differ from normal-weight individuals.

After taking a fasting blood sample, the study participants receive one of the study drinks and a light breakfast. Both should be consumed within 15 minutes. Further blood samples are taken 1, 2, 3, 4 and 6 hours after the drinks have been consumed. To assess the effect of Xanthohumol and Iso-alpha Acids or a combination of both, clinical parameters, blood lipids, blood glucose, uric acid and inflammatory markers will be determined. Furthermore, blood cells, isolated from blood samples of each time point, will be stimulated for measuring inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 - 29,9 kg/m²

as well as one or more of the following incipient metabolic diseases:

* pre-diabetes (fasting blood glucose 100-125 mg/dL),
* fatty liver (grade 1-3),
* high-normal blood pressure to mild hypertension (grade 1, systolic 140-159 mmHg)

Exclusion Criteria:

* History of diseases that could falsify the study results
* inflammatory bowel diseases
* malignant diseases of the gastrointestinal tract
* food allergies
* malabsorption
* kidney or liver disease (except simple fatty liver)
* symptomatic heart failure
* Taking medication to treat these diseases
* Consumption of special diets (e.g. vegan, gluten-free)
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in parameters of immune response | 6 hours
  Changes in concentration of interleukin 6 (ng/ml) in cell culture supernatant of stimulated cells
Changes in parameters of immune response | 6 hours
  Changes in concentrations of interleukin 1 beta (ng/ml) in cell culture supernatant of stimulated cells
Changes in parameters of immune response | 6 hours
  Changes in concentration of tumor necrosis factor alpha (ng/ml) in cell culture supernatant of stimulated cells

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No